CLINICAL TRIAL: NCT00943670
Title: A Phase II, Open-Label Study to Evaluate Corrected QT Interval Effects of Trastuzumab-MCC-DM1 (T-DM1) in Patients With HER2-Positive Locally Advanced or Metastatic Breast Cancer and to Evaluate the Safety and Tolerability of Combined T-DM1 and Pertuzumab in Patients With Early Disease Progression While Receiving T-DM1 Alone
Brief Title: Corrected QT Interval Effects of Trastuzumab Emtansine (T-DM1) in Patients With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Locally Advanced or Metastatic Breast Cancer and the Safety and Tolerability of Combined T-DM1 and Pertuzumab in Patients With Early Disease Progression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDM4688g
Record Dates: First submitted 2009-07-19; First posted 2009-07-22 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Metastatic Breast Cancer
Keywords: MBC; TDM1; Armed Herceptin; Herceptin; Trastuzumab emtansine
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Ado-Trastuzumab Emtansine

ARMS (1):
- T-DM1 / T-DM1 + pertuzumab (Experimental): Trastuzumab emtansine (T-DM1) was administered to participants by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
  From Cycle 4, participants with early progressive disease (demonstrated prior to the end of Cycle 6) could receive combined pertuzumab and trastuzumab emtansine. Pertuzumab was administered after trastuzumab emtansine by IV infusion at a loading dose of 840 mg on Day 1, starting at the cycle after tumor progression was determined, followed by 420 mg IV infusion every 3 weeks in subsequent cycles.
  Participants who met criteria for ongoing clinical benefit were allowed to continue study treatment in the absence of disease progression or unacceptable toxicity for up to 1 year.
  Interventions: Biological: pertuzumab; Biological: Trastuzumab emtansine [Kadcyla]

INTERVENTIONS:
Biological: pertuzumab — Intravenous repeating dose
  Other Names: PERJETA™
Biological: Trastuzumab emtansine [Kadcyla] — Intravenous repeating dose
  Other Names: trastuzumab-MCC-DM1; T-DM1

SUMMARY:
This is a multicenter, open-label, single-arm Phase II study designed to evaluate the effect of T-DM1 on the duration of corrected QT (QTc) interval in patients with HER2-positive locally advanced or metastatic breast cancer and to make preliminary assessments regarding the safety, tolerability, and efficacy of combined T-DM1 and pertuzumab in patients with early disease progression.

The QT interval is a measure of time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. The QTcF interval is the QT interval as calculated using Fridericia's correction; the QTcB interval is the QT interval as calculated using Bazett's correction.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, locally advanced, or metastatic breast cancer; measurable and/or non-measureable but evaluable disease is permitted
* HER2-positive disease
* History of prior trastuzumab therapy
* Life expectancy ≥ 90 days as assessed by the investigator
* Negative urine pregnancy test ≤ 72 hours prior to Cycle 1 Day 1 for all women of childbearing potential
* For patients of childbearing potential, agreement to use one highly effective form of contraception or two effective forms of contraception for the duration of the study treatment(s) and for 4 months after the last dose of T-DM1 or 6 months after the last dose of pertuzumab, if applicable

Exclusion Criteria:

* Any chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or biologic therapy for the treatment of breast cancer within 2 weeks of the first study treatment
* Prior T-DM1 or pertuzumab therapy
* History of intolerance (such as Grade 3-4 infusion reaction) and/or adverse events related to trastuzumab
* Grade ≥ 2 (based on National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v3) peripheral neuropathy at the time of or within 3 weeks prior to the first study treatment
* Brain metastases that are untreated or progressive or have required any type of therapy, including radiation, surgery, and/or steroids, to control symptoms from brain metastases within 60 days prior to the first study treatment
* History of cardiac disease, unstable angina, symptomatic congestive heart failure (CHF) (Class ≥ II per the New York Heart Associate [NYHA] guidelines), myocardial infarction, or ventricular arrhythmia ≤ 6 months prior to Cycle 1, Day 1
* Implantable pacemaker or automatic implantable cardioverter defibrillator
* Congenital long QT syndrome or family history of long QT syndrome
* Current uncontrolled hypertension
* Current treatment with medications that alter cardiac conduction (e.g., digitalis, beta-blockers, or calcium channel blockers) or medications that are generally accepted to have a risk of causing torsades de pointes (TdP)
* Current known active infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus
* Major surgical procedure or significant traumatic injury within 28 days prior to first study treatment, or anticipation of the need for major surgery during the course of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Olsen, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 14 July 2009 and 4 December 2009, 51 patients from 13 study sites in the United States were enrolled and initiated treatment in the study.
Pre-assignment Details: All patients enrolled in the study were initially treated with single-agent trastuzumab emtansine. Participants with early progressive disease could elect to receive pertuzumab in combination with trastuzumab emtansine.
Period: Single-agent Trastuzumab Emtansine
Arm/Group | T-DM1 / T-DM1 + Pertuzumab
Started | 51
Treated | 51
Completed | 9 (Completed single-agent treatment defined as receiving 17 cycles of trastuzumab emtansine therapy.)
Not Completed | 42
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — Systemic progression | 15
Not completed — Adverse Event | 2
Not completed — Early progressive disease | 20
Period: Trastuzumab Emtansine + Pertuzumab
Arm/Group | T-DM1 / T-DM1 + Pertuzumab
Started | 20 (Patients with early progressive disease who elected to receive T-DM1 and pertuzumab.)
Completed | 2 (Completed treatment defined as receiving a total of 17 cycles of therapy in both treatment periods.)
Not Completed | 18
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 4
Not completed — Systemic progression | 6
Not completed — Progression of brain metastases | 2
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | T-DM1 / T-DM1 + Pertuzumab
Number analyzed (Participants) | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 53.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Duration of the QTc Interval
Description: The QT interval is a measure of time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. The corrected QT interval was calculated using Fridericia's correction (QTcF) from electrocardiogram (ECG) data. Each participant had triplicate QTcF intervals measured at each timepoint and the average was calculated for each patient at each timepoint. For each timepoint, a participant's corresponding baseline QTcF interval was subtracted from the average QTcF intervals to create a baseline-adjusted average QTcF interval.
Time Frame: Cycle 1 Day 1, pre-dose (Baseline); Cycle 1 Day 1, 15 and 60 minutes post-dose; Cycle 1 Day 8; and Cycle 3 Day 1, 15 minutes pre-dose and 15 and 60 minutes post-dose.
Population: ECG-evaluable population consisted of patients who received T-DM1, had at least 1 interpretable pre-T-DM1 ECG measurement recorded on Cycle 1 Day 1, had at least 1 interpretable post-T-DM1 ECG measurement and who were not treated with medications that may have altered cardiac conduction. N indicates the ECG-evaluable population at each time point.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- T-DM1: Trastuzumab emtansine (T-DM1) was administered to participants by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
Arm/Group | T-DM1
Number analyzed (Participants) | 51
milliseconds
  Cycle 1, Day 1, 15 minutes post-dose [N=44] | 1.2 (8.3)
  Cycle 1, Day 1, 60 minutes post-dose [N=45] | -1.0 (6.3)
  Cycle 1, Day 8 [N=43] | -4.0 (13.4)
  Cycle 3, Day 1, 15 minutes pre-dose [N=35] | -0.1 (10.1)
  Cycle 3, Day 1, 15 minutes post-dose [N=37] | 4.7 (9.6)
  Cycle 3, Day 1, 60 minutes post-dose [N=37] | 4.7 (10.9)

2. Secondary Outcome: Change From Baseline in Mean Duration of the QTc Interval Using Bazett's Correction
Description: The corrected QT interval was calculated using Bazett's correction (QTcB) from electrocardiogram (ECG) data. Each participant had triplicate QTcB intervals measured at each timepoint and the average was calculated for each patient at each timepoint. For each timepoint, a participant's corresponding baseline QTcB interval was subtracted from the average QTcB intervals to create a baseline-adjusted average QTcB interval.
Time Frame: as for outcome 1
Population: ECG-Evaluable population; N indicates the ECG-evaluable population with available data at each time point.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | T-DM1
Number analyzed (Participants) | 51
milliseconds
  Cycle 1, Day 1, 15 minutes post-dose [N=44] | 3.6 (9.1)
  Cycle 1, Day 1, 60 minutes post-dose [N=45] | 2.6 (7.4)
  Cycle 1, Day 8 [N=43] | 0.7 (13.1)
  Cycle 3, Day 1, 15 minutes pre-dose [N=35] | 3.7 (14.5)
  Cycle 3, Day 1, 15 minutes post-dose [N=37] | 6.0 (13.2)
  Cycle 3, Day 1, 60 minutes post-dose [N=37] | 7.3 (12.2)

3. Secondary Outcome: Change From Baseline in Uncorrected QT Interval
Description: The uncorrected QT interval was calculated from electrocardiogram (ECG) data. Each participant had triplicate QT intervals measured at each timepoint and the average was calculated for each patient at each timepoint. For each timepoint, a participant's corresponding baseline QT interval was subtracted from the average QT intervals to create a baseline-adjusted average QT interval.
Time Frame: as for outcome 1
Population: ECG-Evaluable population; N indicates the ECG-evaluable population with available data at each time point.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | T-DM1
Number analyzed (Participants) | 51
milliseconds
  Cycle 1 Day 1, 15 minutes post-dose [N=44] | -2.6 (17.4)
  Cycle 1 Day 1, 60 minutes post-dose [N=45] | -7.0 (14.9)
  Cycle 1 Day 8 [N=43] | 12.2 (22.1)
  Cycle 3 Day 1, 15 minutes pre-dose [N=35] | -7.0 (14.9)
  Cycle 3 Day 1, 15 minutes post-dose [N=37] | 2.4 (16.4)
  Cycle 3 Day 1, 60 minutes post-dose [N=37] | 0.1 (19.6)

4. Secondary Outcome: Change From Baseline in PR Interval
Description: The PR interval is the time in seconds from the beginning of the P wave to the beginning of the QRS complex, and was calculated from electrocardiogram (ECG) data. Each participant had triplicate PR intervals measured at each timepoint and the average was calculated for each patient at each timepoint. For each timepoint, a participant's corresponding baseline PR interval was subtracted from the average PR intervals to create a baseline-adjusted average PR interval.
Time Frame: as for outcome 1
Population: ECG-Evaluable population
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | T-DM1
Number analyzed (Participants) | 51
milliseconds
  Cycle 1 Day 1, 15 minutes post-dose [N=44] | 2.3 (7.5)
  Cycle 1 Day 1, 60 minutes post-dose [N=45] | 2.5 (8.7)
  Cycle 1 Day 8 [N=43] | -0.7 (10.7)
  Cycle 3 Day 1, 15 minutes pre-dose [N=35] | 1.8 (11.0)
  Cycle 3 Day 1, 15 minutes post-dose [N=37] | 6.7 (9.8)
  Cycle 3 Day 1, 60 minutes post-dose [N=37] | 5.3 (8.6)

5. Secondary Outcome: Change From Baseline in QRS Duration
Description: The QRS interval represents the time it takes for depolarization of the ventricles and was calculated from electrocardiogram (ECG) data. Each participant had triplicate QRS intervals measured at each timepoint and the average was calculated for each patient at each timepoint. For each timepoint, a participant's corresponding baseline QRS interval was subtracted from the average QRS intervals to create a baseline-adjusted average QRS interval.
Time Frame: as for outcome 1
Population: ECG-Evaluable population; N indicates the ECG-evaluable population with available data at each time point.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | T-DM1
Number analyzed (Participants) | 51
milliseconds
  Cycle 1 Day 1, 15 minutes post-dose [N=44] | 1.2 (3.1)
  Cycle 1 Day 1, 60 minutes post-dose [N=45] | 0.4 (3.0)
  Cycle 1 Day 8 [N=43] | 1.1 (4.8)
  Cycle 3 Day 1, 15 minutes pre-dose [N=35] | 0.5 (4.5)
  Cycle 3 Day 1, 15 minutes post-dose [N=37] | 1.9 (4.0)
  Cycle 3 Day 1, 60 minutes post-dose [N=37] | 1.5 (3.8)

6. Secondary Outcome: Change From Baseline in Heart Rate
Time Frame: as for outcome 1
Population: ECG-evaluable population; N indicates the ECG-evaluable population with available data at each time point.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | T-DM1
Number analyzed (Participants) | 51
beats per minute
  Cycle 1 Day 1, 15 minutes post-dose [N=44] | 2.9 (8.3)
  Cycle 1 Day 1, 60 minutes post-dose [N=45] | 4.4 (7.9)
  Cycle 1 Day 8 [N=43] | 5.4 (8.8)
  Cycle 3 Day 1, 15 minutes pre-dose [N=35] | 4.1 (7.9)
  Cycle 3 Day 1, 15 minutes post-dose [N=37] | 0.8 (7.6)
  Cycle 3 Day 1, 60 minutes post-dose [N=37] | 2.4 (7.8)

7. Secondary Outcome: Percentage of Participants Within Each Absolute QTc Interval Category
Description: The corrected QT interval was calculated using Fridericia's correction (QTcF) and using Bazett's correction (QTcB) from electrocardiogram (ECG) data. Each participant had triplicate QTc intervals measured at each timepoint and the average was calculated for each patient at each timepoint. QTc interval categories are based off International Conference on Harmonisation (ICH) Tripartite Guideline E14.
Time Frame: Cycle 1 Day 1, 15 and 60 minutes post-dose; Cycle 1 Day 8; and Cycle 3 Day 1, 15 minutes pre-dose and 15 and 60 minutes post-dose.
Population: The number of participants analyzed for each QTc interval category represents the total treated population. N indicates the ECG-evaluable population with available data at each time point.
Measure: Number; unit: percentage of participants
Groups:
- Average QTc Interval ≤ 450 ms: Participants with an average QTc interval less than or equal to 450 ms who received trastuzumab emtansine (T-DM1) by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
- Average QTc Interval > 450 to ≤ 480 ms: Participants with an average QTc interval greater than 450 and less than or equal to 480 ms who received trastuzumab emtansine (T-DM1) by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
- Average QTc Interval > 480 to ≤ 500 ms: Participants with an average QTc interval greater than 480 and less than or equal to 500 ms who received trastuzumab emtansine (T-DM1) by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
- Average QTc Interval > 500 ms: Participants with an average QTc interval greater than 500 ms who received trastuzumab emtansine (T-DM1) by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
Arm/Group | Average QTc Interval ≤ 450 ms | Average QTc Interval > 450 to ≤ 480 ms | Average QTc Interval > 480 to ≤ 500 ms | Average QTc Interval > 500 ms
Number analyzed (Participants) | 51 | 51 | 51 | 51
percentage of participants
  QTcF: Cycle 1, Day 1, 15 minutes post-dose [N=44] | 100 | 0 | 0 | 0
  QTcF: Cycle 1, Day 1, 60 minutes post-dose [N=45] | 100 | 0 | 0 | 0
  QTcF: Cycle 1, Day 8 [N=43] | 100 | 0 | 0 | 0
  QTcF: Cycle 3, Day 1, 15 minutes pre-dose [N=35] | 97.1 | 2.9 | 0 | 0
  QTcF: Cycle 3, Day 1, 15 minutes post-dose [N=37] | 94.6 | 5.4 | 0 | 0
  QTcF: Cycle 3, Day 1, 60 minutes post-dose [N=37] | 97.3 | 2.7 | 0 | 0
  QTcB: Cycle 1, Day 1, 15 minutes post-dose [N=44] | 79.5 | 20.5 | 0 | 0
  QTcB: Cycle 1, Day 1, 60 minutes post-dose [N=45] | 73.3 | 26.7 | 0 | 0
  QTcB: Cycle 1, Day 8 [N=43] | 79.1 | 20.9 | 0 | 0
  QTcB: Cycle 3, Day 1, 15 minutes pre-dose [N=35] | 82.9 | 17.1 | 0 | 0
  QTcB: Cycle 3, Day 1, 15 minutes post-dose [N=37] | 70.3 | 29.7 | 0 | 0
  QTcB: Cycle 3, Day 1, 60 minutes post-dose [N=37] | 70.3 | 29.7 | 0 | 0

8. Secondary Outcome: Percentage of Participants Within Each Baseline-adjusted QTc Interval Category
Description: The corrected QT interval was calculated using Fridericia's correction (QTcF) and using Bazett's correction (QTcB) from electrocardiogram (ECG) data. Each participant had triplicate QTc intervals measured at each timepoint and the average was calculated for each patient at each timepoint. For each timepoint, a participant's corresponding baseline QTc interval was subtracted from the average QTc intervals to create a baseline-adjusted average QTc interval.
  QTc interval categories are based off International Conference on Harmonisation (ICH) Tripartite Guideline E14.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Groups:
- Baseline-adjusted QTc Interval ≤ 30 ms: Participants with an average Baseline-adjusted QTc interval less than or equal to 30 ms who received trastuzumab emtansine (T-DM1) by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
- Baseline-adjusted QTc Interval > 30 to ≤ 60 ms: Participants with an average Baseline-adjusted QTc interval greater than 30 and less than or equal to 60 ms who received trastuzumab emtansine (T-DM1) by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
- Baseline-adjusted QTc Interval > 60 ms: Participants with an average Baseline-adjusted QTc interval greater than 60 ms who received trastuzumab emtansine (T-DM1) by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
Arm/Group | Baseline-adjusted QTc Interval ≤ 30 ms | Baseline-adjusted QTc Interval > 30 to ≤ 60 ms | Baseline-adjusted QTc Interval > 60 ms
Number analyzed (Participants) | 51 | 51 | 51
percentage of participants
  QTcF: Cycle 1, Day 1, 15 minutes post-dose [N=44] | 100 | 0 | 0
  QTcF: Cycle 1, Day 1, 60 minutes post-dose [N=45] | 100 | 0 | 0
  QTcF: Cycle 1, Day 8 [N=43] | 100 | 0 | 0
  QTcF: Cycle 3, Day 1, 15 minutes pre-dose [N=35] | 100 | 0 | 0
  QTcF: Cycle 3, Day 1, 15 minutes post-dose [N=37] | 100 | 0 | 0
  QTcF: Cycle 3, Day 1, 60 minutes post-dose [N=37] | 100 | 0 | 0
  QTcB: Cycle 1, Day 1, 15 minutes post-dose [N=44] | 100 | 0 | 0
  QTcB: Cycle 1, Day 1, 60 minutes post-dose [N=45] | 100 | 0 | 0
  QTcB: Cycle 1, Day 8 [N=43] | 100 | 0 | 0
  QTcB: Cycle 3, Day 1, 15 minutes pre-dose [N=35] | 94.3 | 5.7 | 0
  QTcB: Cycle 3, Day 1, 15 minutes post-dose [N=37] | 94.6 | 5.4 | 0
  QTcB: Cycle 3, Day 1, 60 minutes post-dose [N=37] | 97.3 | 2.7 | 0

9. Secondary Outcome: Percentage of Participants With New Abnormal U Waves
Description: The incidence of abnormal U-wave changes from baseline was determined based on centrally read electrocardiogram (ECG) tracings comparing each of the three triplicate readings from the post baseline ECG time points to the baseline ECG reading. At each time point, if at least one of the three triplicate readings was abnormal, the participant was counted as abnormal for that ECG timepoint as follows: a large U wave, inverted U wave, or T-U fusion compared with baseline was considered an abnormal significant change from baseline.
Time Frame: as for outcome 1
Population: ECG-evaluable population; N indicates the ECG-evaluable population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | T-DM1
Number analyzed (Participants) | 51
percentage of participants
  Cycle 1, Day 1, 15 minutes post-dose [N=44] | 0
  Cycle 1, Day 1, 60 minutes post-dose [N=45] | 0
  Cycle 1, Day 8 [N=43] | 0
  Cycle 3, Day 1, 15 minutes pre-dose [N=35] | 0
  Cycle 3, Day 1, 15 minutes post-dose [N=36] | 0
  Cycle 3, Day 1, 60 minutes post-dose [N=37] | 0

10. Secondary Outcome: Percentage of Participants With New Abnormal T Waves
Description: The incidence of abnormal T-wave changes from baseline was determined based on centrally read electrocardiogram (ECG) tracings comparing each of the three triplicate readings from the post baseline ECG time points to the baseline ECG reading. At each time point, if at least one of the three triplicate readings was abnormal, the participant was counted as abnormal for that ECG timepoint as follows: an inverted T, flat T, or biphasic T compared with baseline was considered an abnormal significant change from baseline. Additionally, nonspecific T-wave changes from baseline were considered as abnormal nonsignificant changes from baseline. T-wave changes from baseline due to ventricular conduction or left ventricular hypertrophy strain were considered not evaluable. C=Cycle; D=Day.
Time Frame: as for outcome 1
Population: ECG-Evaluable population; N indicates the ECG-evaluable population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | T-DM1
Number analyzed (Participants) | 51
percentage of participants
  Significant: C1D1, 15 minutes post-dose [N=44] | 0
  Significant: C1D1, 60 minutes post-dose [N=45] | 0
  Significant: C1D8 [N=43] | 2.3
  Significant: C3D1, 15 minutes pre-dose [N=35] | 0
  Significant: C3D1, 15 minutes post-dose [N=36] | 0
  Significant: C3D1, 60 minutes post-dose [N=37] | 0
  Non-Significant: C1D1, 15 minutes post-dose [N=44] | 13.6
  Non-Significant: C1D1, 60 minutes post-dose [N=45] | 11.1
  Non-Significant: C1D8 [N=43] | 20.9
  Non-Significant: C3D1, 15 minutes pre-dose [N=35] | 17.1
  Non-Significant: C3D1, 15 minutes post-dose [N=36] | 13.9
  Non-Significant: C3D1, 60 minutes post-dose [N=37] | 27.0

11. Secondary Outcome: Percentage of Participants With an Objective Response During the Single-agent Trastuzumab Emtansine Treatment Period
Description: Objective response was defined as a complete response (CR) or partial response (PR) determined on two consecutive assessments conducted by the investigator ≥ 4 weeks apart. Responses were assessed by physical examination and imaged-based evaluation using a modified version of the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0:
  CR-the disappearance of all target lesions and the disappearance of all nontarget lesions and normalization of tumor marker level and no new lesions.
  PR-either the disappearance of all target lesions with persistence of one or more nontarget lesion(s) and/or the maintenance of tumor marker level above the normal limits, or, at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter with no new lesions or unequivocal progression of existing nontarget lesions.
Time Frame: Tumor assessments were performed after every three cycles until study termination or progressive disease (up to a maximum of one year).
Population: The efficacy-evaluable population was defined as patients who received at least one dose of study drug. Patients with missing or no post-baseline response assessments were classified as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- T-DM1: Trastuzumab emtansine (T-DM1) was administered to participants by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
  Participants who met criteria for ongoing clinical benefit were allowed to continue study treatment in the absence of disease progression or unacceptable toxicity for up to 1 year.
Arm/Group | T-DM1
Number analyzed (Participants) | 51
percentage of participants | 25.5 [15.2 to 38.5]

12. Secondary Outcome: Duration of Objective Response Based on Investigator Assessment During the Single-agent Trastuzumab Emtansine Treatment Period
Description: In patients with an objective response during the single-agent trastuzumab emtansine treatment period, duration of response was defined as the time from the first documented objective response to the time of first documented disease progression or death, whichever occurred first. Progressive disease was defined as either at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study with an absolute increase of at least 5 mm, or the appearance of one or more new lesions, or the unequivocal progression of existing nontarget lesions.
  If a patient did not die or experience disease progression before the end of the study, duration of response was censored at the day of the last tumor assessment when the patient was known to be progression free.
Time Frame: Time from the first documented objective response to the time of first documented disease progression or death, up to a maximum time period of one year.
Population: Efficacy evaluable patients who achieved an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DM1
Number analyzed (Participants) | 13
months | 9.3 [4.7 to NA] — Upper limit of the confidence not estimable due to the low number of patients with an event (7).

13. Secondary Outcome: Progression-free Survival During the Single-agent Trastuzumab Emtansine Treatment Period
Description: Progression-free survival (PFS) was defined as the time from the first day of study treatment (Day 1) to first documented disease progression or death, whichever occurred first. If a patient did not experience disease progression or die, PFS was censored at the day of the last tumor assessment that a patient was known to be progression free.
Time Frame: From the first day of study treatment to the first documented disease progression or death, up to a maximum time period of one year.
Population: Efficacy evaluable patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DM1
Number analyzed (Participants) | 51
months | 4.3 [4.0 to 6.7]

14. Secondary Outcome: Percentage of Participants With Clinical Benefit During the Single-agent Trastuzumab Emtansine Treatment Period
Description: Participants were considered to have experienced clinical benefit if they had an objective response or maintained stable disease for at least 6 months from start of study treatment. Objective response was defined as a complete or partial response determined on two consecutive tumor assessments at least 4 weeks apart based on a modified version of RECIST.
  Stable disease was defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started and no new lesions or unequivocal progression of existing nontarget lesions.
Time Frame: as for outcome 11
Population: The efficacy-evaluable population was defined as patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DM1
Number analyzed (Participants) | 51
percentage of participants | 39.2 [25.8 to 53.1]

15. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An serious AE is any AE that is fatal, life threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product(s), or is considered a significant medical event by the investigator (e.g., may jeopardize the patient or may require medical/surgical intervention to prevent one of the outcomes listed above).
  The severity of each AE was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0, or as follows: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Very severe; Grade 5 = Death related to AE.
Time Frame: From first dose until 30 days after last dose (up to 1 year).
Population: Safety-Evaluable Patients (i.e., the treated population).
Measure: Number; unit: participants
Groups:
- T-DM1 + Pertuzumab: Participants who received combined pertuzumab and trastuzumab emtansine. Pertuzumab was administered after trastuzumab emtansine by IV infusion at a loading dose of 840 mg on Day 1, followed by 420 mg IV infusion every 3 weeks in subsequent cycles.
Arm/Group | T-DM1 | T-DM1 + Pertuzumab
Number analyzed (Participants) | 51 | 20
participants
  Any adverse event | 51 | 18
  Grade ≥ 3 adverse events | 17 | 12
  Serious adverse events | 4 | 5
  Adverse events leading to treatment discontinuatio | 2 | 5
  Deaths | 0 | 0

16. Secondary Outcome: Number of Participants With Decreased Ejection Fraction
Description: Left ventricular ejection fraction (LVEF) was assessed on the basis of local assessments of echocardiogram or multigated acquisition scan (MUGA) data. A decrease in LVEF is defined as a decrease from Baseline of greater than or equal to 15%.
  Grade 3 LVEF is an ejection fraction between 20 and 40%.
Time Frame: Assessed at Baseline and after every 3 cycles, up to 1 year.
Population: Safety-Evaluable Patients (i.e., the treated population).
Measure: Number; unit: participants
Arm/Group | T-DM1 | T-DM1 + Pertuzumab
Number analyzed (Participants) | 51 | 20
participants
  Grade 3 | 1 | 0
  Overall | 1 | 1

17. Secondary Outcome: Maximum Observed Serum Concentration of T-DM1 and Total Trastuzumab
Description: Serum samples were quantitated for T-DM1 (DM1 conjugated to trastuzumab) levels in a validated assay using an indirect sandwich enzyme-linked immunosorbent assay (ELISA). The minimum quantifiable concentration in human serum was 40 ng/mL. Serum samples were assayed for total trastuzumab (conjugated and unconjugated T-DM1) in a validated assay using an indirect sandwich ELISA method; the minimum quantifiable concentration in human serum was 40 ng/mL.
Time Frame: Blood samples were collected prior to dosing, 15 and 60 minutes after the end of infusion, and anytime on Days 8 and 15 in Cycles 1 and 3, and pre-dose in Cycle 4.
Population: Pharmacokinetic (PK)-evaluable patients were defined as patients who had adequate concentration-time data to estimate at least one PK parameter. "N" refers to the number of PK-evaluable patients in that cycle.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Single-Agent T-DM1 Treatment: Trastuzumab emtansine (T-DM1) was administered to participants by intravenous (IV) infusion on Day 1 of every 3 week cycle at a dose of 3.6 mg/kg.
Arm/Group | Single-Agent T-DM1 Treatment
Number analyzed (Participants) | 51
μg/mL
  Cycle 1: T-DM1 [N=51] | 75.6 (21.9)
  Cycle 1: Total trastuzumab [N=51] | 95.9 (32.3)
  Cycle 3: T-Dm1 [N=47] | 80.7 (18.1)
  Cycle 3: Total trastuzumab [N=47] | 98.6 (26.1)

18. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Time of Last Measurable Concentration for T-DM1 and Total Trastuzumab
Description: Area under the serum concentration-time curve from Time zero to time of last measurable concentration (AUClast) for T-DM1 (conjugated trastuzumab) and Total Trastuzumab (conjugated and unconjugated T-DM1) at Cycle 1 and Cycle 3.
Time Frame: Blood samples were collected prior to T-DM1 dosing, 15 and 60 minutes after the end of infusion, and anytime on Days 8 and 15 in Cycles 1 and 3, and pre-dose in Cycle 4.
Population: PK-evaluable patients were defined as patients who had adequate concentration-time data to estimate at least one PK parameter. "N" refers to the number of PK-evaluable patients in that cycle.
Measure: Mean (Standard Deviation); unit: μg * day/mL
Arm/Group | Single-Agent T-DM1 Treatment
Number analyzed (Participants) | 51
μg * day/mL
  Cycle 1: T-DM1 [N=51] | 418 (121)
  Cycle 1: Total trastuzumab [N=51] | 929 (564)
  Cycle 3: T-Dm1 [N=47] | 475 (150)
  Cycle 3: Total trastuzumab [N=47] | 958 (394)

19. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity for T-DM1 and Total Trastuzumab
Description: Area under the serum concentration-time curve from Time zero extrapolated to infinity (AUCinf) for T-DM1 (conjugated trastuzumab) and total trastuzumab (conjugated and unconjugated T-DM1) at Cycle 1.
Time Frame: Blood samples were collected prior to T-DM1 dosing, 15 and 60 minutes after the end of infusion, and anytime on Days 8 and 15 in Cycle 1.
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: μg * day/mL
Arm/Group | Single-Agent T-DM1 Treatment
Number analyzed (Participants) | 51
μg * day/mL
  T-DM1 | 431 (126)
  Total trastuzumab | 1420 (1390)

20. Secondary Outcome: Terminal Half-life for T-DM1 and Total Trastuzumab
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Single-Agent T-DM1 Treatment
Number analyzed (Participants) | 51
days
  Cycle 1: T-DM1 [N=51] | 4.02 (0.938)
  Cycle 1: Total trastuzumab [N=51] | 10.3 (6.81)
  Cycle 3: T-Dm1 [N=47] | 4.46 (0.926)
  Cycle 3: Total trastuzumab [N=47] | 12.0 (6.24)

21. Secondary Outcome: Clearance T-DM1 and Total Trastuzumab
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Single-Agent T-DM1 Treatment
Number analyzed (Participants) | 51
mL/day/kg
  Cycle 1: T-DM1 [N=51] | 9.17 (3.03)
  Cycle 1: Total trastuzumab [N=51] | 4.21 (2.43)
  Cycle 3: T-Dm1 [N=47] | 7.91 (3.30)
  Cycle 3: Total trastuzumab [N=47] | 3.12 (1.71)

22. Secondary Outcome: Volume of Distribution at Steady State for T-DM1 and Total Trastuzumab
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Single-Agent T-DM1 Treatment
Number analyzed (Participants) | 51
mL/kg
  Cycle 1: T-DM1 [N=51] | 41.2 (24.5)
  Cycle 1: Total trastuzumab [N=51] | 41.9 (16.2)
  Cycle 3: T-Dm1 [N=47] | 43.6 (40.7)
  Cycle 3: Total trastuzumab [N=47] | 43.7 (15.4)

23. Secondary Outcome: Number of Participants With Anti-therapeutic Antibodies (ATAs) to Trastuzumab Emtansine
Description: The number of participants with anti-T-DM1 antibodies was assessed using a validated bridging antibody enzyme-linked immunosorbent assay (ELISA).
Time Frame: as for outcome 18
Population: Evaluable patients, defined as patients who had at least one ATA measurement available for analysis at Baseline (pre-dose in Cycle 1) and post-baseline.
Measure: Number; unit: participants
Arm/Group | Single-Agent T-DM1 Treatment
Number analyzed (Participants) | 47
participants
  Pre-dose (Baseline) | 2
  Post-dose | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Single-Agent T-DM1 Treatment | T-DM1 + Pertuzumab
Serious Adverse Events (participants affected / at risk) | 4/51 | 5/20
Other Adverse Events (participants affected / at risk) | 51/51 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Agent T-DM1 Treatment (N=51) | T-DM1 + Pertuzumab (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Agent T-DM1 Treatment (N=51) | T-DM1 + Pertuzumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0
Cardiac flutter (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 4 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 6 | 1
Vomiting (Gastrointestinal disorders) | 16 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 33 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Dry mouth (Gastrointestinal disorders) | 25 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 12 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 33 | 4
Pain (General disorders) | 4 | 4
Pyrexia (General disorders) | 12 | 2
Catheter site erythema (General disorders) | 0 | 1
Chest discomfort (General disorders) | 2 | 1
Chest pain (General disorders) | 1 | 1
Drug effect increased (General disorders) | 0 | 1
Medical device complication (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Thirst (General disorders) | 1 | 1
Chills (General disorders) | 11 | 0
Asthenia (General disorders) | 3 | 0
Gait disturbance (General disorders) | 3 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 3
Catheter site cellulitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 9 | 0
Herpes zoster (Infections and infestations) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 17 | 4
Blood alkaline phosphatase increased (Investigations) | 4 | 4
Alanine aminotransferase increased (Investigations) | 7 | 2
Weight decreased (Investigations) | 5 | 2
Ejection fraction decreased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 1
International normalised ratio increased (Investigations) | 0 | 1
Weight increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 8 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dizziness (Nervous system disorders) | 5 | 2
Headache (Nervous system disorders) | 11 | 2
Ataxia (Nervous system disorders) | 1 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 6 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 1
Sedation (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 6 | 0
Paraesthesia (Nervous system disorders) | 5 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 0
Depression (Psychiatric disorders) | 3 | 3
Anxiety (Psychiatric disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 8 | 2
Food aversion (Psychiatric disorders) | 0 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 6 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 4 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 0
Flushing (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.